CLINICAL TRIAL: NCT02295254
Title: Microbiome Changes in Travelers to Tropical Destinations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Prof. Eli Schwartz MD, DTMH, Principal Investigator of geographic clinic, Sheba Medical Center
Other Study IDs: SHEBA-14-1543-ES-CTIL
Record Dates: First submitted 2014-11-11; First posted 2014-11-20 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Intestinal Diseases
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Research group: The study contain only one group: travelers who intended to travel to tropical destinations. The participants will give a feces sample before and after the travel.
  Interventions: Other: feces sample

INTERVENTIONS:
Other: feces sample — The travelers will give feces sample before and after the travel. The sample microorganisms will be analyzed.

SUMMARY:
The human gut contain a wide range of microorganisms creating the gut microbiome. The microbiome has great impact on metabolic and immunologic processes and responses. Travelers who travel to tropical destinations where the intestinal infection risk is high are prone to microbiome changes. During the current study the travelers will give feces specimen before and after the travel and their microbiome will be analyzed.

DETAILED DESCRIPTION:
Individual differences in the microorganisms variety are affected by external factors such as food, age, geographic location, medication consumption, host genetics and exposure to microorganisms in early stages of life. During the current study the geographic location affect will be tested by comparing the microorganism environment before and after traveling to tropical destinations.

ELIGIBILITY:
Inclusion Criteria:

* Travelers who intended to travel to tropical areas
* Good general health

Exclusion Criteria:

* Medication consumption
* Background diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Travelers who intended to travel to tropical areas.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Type and number of intestinal microorganisms | 1 year
  The participants microbiome will be analyzed before and after the travel. The type and number of microorganisms will be determined by microbiological measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Schwartz, MD, DTMH, Principal Investigator — Eli.schwartz@sheba.health.gov.il
Locations (1):
- Center of Geographic Medicine, Tel Litwinsky, Israel